CLINICAL TRIAL: NCT00683527
Title: New Versus Standard Enteral Iron Supplementation Regime in Very Low Birth Weight Infants - A Randomized Controlled Trial
Brief Title: Timing of Iron Supplementation in Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: M Jeeva Sankar, Department of Pediatrics, AIIMS, New Delhi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A-34/2006
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Nutritional Status
Keywords: Iron supplementation; Timing; Serum ferritin; Very low birth weight infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Starting oral iron at day 14 of life (Early Iron group)
  Interventions: Drug: Elemental iron
- 2 (No Intervention): No iron supplementation till 60 days of life (Control group)

INTERVENTIONS:
Drug: Elemental iron — Iron in the dose of 3-4 mg/kg/day (of elemental iron) PO once daily mixed with expressed breast milk from 14 days of life till the end of study period
  Other Names: 'Tonoferon' drops, East India Co
  Arms: 1

SUMMARY:
To examine if early iron supplementation (starting oral iron at 14 days of life) would improve the nutritional iron status(measured by serum ferritin) of very low birth weight infants at postnatal age of 60 days, when compared to the standard regime of starting iron at 2 months of life.

DETAILED DESCRIPTION:
Smaller the preterm infants at birth, more susceptible they are to iron deficiency due to low body iron stores. Despite having low iron stores, very low birth weight (VLBW) infants are not usually started on iron supplementation till they reach a postnatal age of 6 to 8 weeks. Such delayed supplementation can lead to rapid depletion of iron stores when erythropoiesis becomes active (by 8 weeks of life).

Depletion of iron stores is the first step in the continuum of changes that occur in iron deficiency. Iron deficiency induces biochemical defects (such as impaired synthesis of DNA and collagen) even before any features of microcytic, hypochromic anemia become evident. The rapidly maturing preterm brain is especially vulnerable to the effects of iron deficiency; poor school-age performance has been reported among children who had low iron stores in their neonatal period.

Early iron supplementation i.e. starting iron once the infant reaches full enteral feeds could potentially improve the iron stores and prevent its depletion. Surprisingly, few studies are available till date to support (or refute!) this view. The current study was designed to test the hypothesis whether early iron supplementation would increase the nutritional iron status (as measured by serum ferritin) at 60 days of life when compared to the existing regime of starting iron at the age 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Infants who have reached at least 100 ml/kg/day of oral feeds by day 14 of life

Exclusion Criteria:

* Major congenital anomalies
* Rh hemolytic disease
* Twin-to-twin transfusion syndrome
* Refusal to give consent

Ages: 14 Days to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2006-05; Primary Completion 2006-11 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Serum ferritin | 60 days postnatal age

SECONDARY OUTCOMES:
Composite outcome of neonatal morbidities that include chronic lung disease [CLD], necrotizing enterocolitis [NEC-any stage], periventricular leucomalacia [PVL], and retinopathy of prematurity [ROP] requiring treatment | Till the end of study period (2 months)
Hematologic and anthropometric parameters | at 60 days of age
Requirement of blood transfusion | till the end of study period

CONTACTS AND LOCATIONS:
Overall Officials: M Jeeva Sankar, MD DM, Principal Investigator — All India Institute of Medical Sciences; Vinod K Paul, MD PhD, Study Chair — All India Institute of Medical Sciences; Ramesh Agarwal, MD DM, Study Chair — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, Delhi (UT), India